CLINICAL TRIAL: NCT04554784
Title: A Prospective Randomized Control Trial on the Effectiveness of Bowen Therapy for Pain Management in Patients With Fibromyalgia
Brief Title: Effectiveness of Bowen Therapy for Pain Management in Patients With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alice Ho Miu Ling Nethersole Hospital (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ms Pik Yu CHEN, Pain nurse (Registered Nurse), Alice Ho Miu Ling Nethersole Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bowen (fibro) 2020.357
Record Dates: First submitted 2020-09-11; First posted 2020-09-18 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Fibromyalgia
Keywords: Bowen Therapy; conventional pain management
MeSH Terms: conditions — Fibromyalgia | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to receive either conventional treatment or Bowen Therapy, following the computer-generated sequence (1= Control, 2= Bowen Therapy). The randomization sequence will be prepared by a research assistant, who will not take part in the study. The randomization sequence will be placed in a brown, and sealed envelopes: Group 1 (n= 40): Control (conventional treatment); and Group 2 (n= 40): Bowen Therapy.
Who Masked: Investigator, Outcomes Assessor
Masking Description: 1. Investigator will be blinded and responsible for obtaining informed consent.
  2. Outcome Assessor who will be responsible to perform the Endurance Strength Test (EST) and assist patients in completing questionnaires, will be blinded to measure the EST during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Conventional pain treatment.
  Interventions: Other: Conventional
- Bowen (Active Comparator): Patients will be referred to Occupational Therapist for Bowen therapy.
  Interventions: Procedure: Bowen

INTERVENTIONS:
Other: Conventional — Patients' condition will be continue managed by pain specialists with regular follow-ups and continue patients' active concurrent pain treatment such as taking analgesics, physiotherapy, massage, chiropractor.
  Arms: Conventional
Procedure: Bowen — Patients will be referred to Occupational therapist for Bowen Therapy. There will be a week washout period before the start of Bowen Therapy. During a week washout period and study period, patients can continue taking analgesia, but advised to stop the concurrent treatments which can affect the deep tissue such as massage, physiotherapy, and chiropractic to minimize the counteracting effect on the Bowen's action.
  During a Bowen Therapy session, patients will lie relaxed on the examination couch wearing loosely fitting clothing or only the affected area being exposed. The therapist applies a series of gentle movements across the body. The gentle movements focus on a body of muscle, tendon or nerve and release tension through the nerve within the area. Each session will last for 30 minutes to an hour. After each session, the next appointment will be given to patients. The first four sessions will be scheduled on weekly basis, and the remaining four on biweekly session.
  Arms: Bowen

SUMMARY:
The aim of this prospective, randomized study is to explore the effectiveness of Bowen Therapy in pain management for patients with fibromyalgia. In Hong Kong, Bowen Therapy is a non-invasive technique and one of the treatment modalities adopted by Occupational Therapists. Bowen Therapy uses specific sequences of gentle cross-fibre moves over muscles, tendons, ligaments, and fascia to stimulate or improve the flow of blood and lymph, and thus activate the body's healing mechanisms that enhances tissue repair. As a result, it can lessen pain and tension, restore more optimal body function, and subsequently alleviate emotional and psychological stress associated with the pain. Bowen Therapy is widely recognized and utilized worldwide for acute and chronic health conditions from new-born to the elderly, both mobilized and bed-ridden patients with no documented evidence to show it has caused any harm or adverse effects.

There are two study groups in this study and patients will be randomized and allocated to either one. One group (Control group) will continue receiving conventional treatment; while another group (Bowen group) will receive 8 sessions of Bowen therapy. The investigators hypothesize that Bowen Therapy is superior to the conventional pain treatment for patients with fibromyalgia.

DETAILED DESCRIPTION:
This study is going to look at the effectiveness of Bowen Therapy in pain management for patients with fibromyalgia. 80 patients with fibromyalgia attending pain management clinic will be recruited at Alice Ho Miu Ling Nethersole Hospital after informed consent. They will be randomized into either group (control group or Bowen group). Control group will continue receiving conventional treatment such as follow-ups by pain specialists, taking analgesia, physiotherapy. Bowen group will need to attend 8 sessions of therapy. All subjects will be evaluated at 12th week and 24th week after signing the consent.

ELIGIBILITY:
Inclusion Criteria:

* Widespread pain index (WPI) ≧7 and symptom severity (SS) scale score ≧5 or WPI between 3 and 6 with SS scale score ≧9. The WPI includes evaluation of tender points at 19 regions. Tender point count (TPC) is examined by application of approximately 4 kg/cm2 pressure with the tip of the thumb on those regions.
* Symptoms have been present at a similar level for at least 3 months.
* Patient does not have any disorder that would otherwise explain the pain
* Agrees to participate in the study and agree to discontinue other alternatives treatments except in conditions otherwise approved by the investigators.

Exclusion Criteria:

* Patient refusal
* pregnancy
* assessed to be contraindicated to participate by pain specialists due to the presence of other co-morbidities or conditions
* underlining disease that affect mobility of upper limb and lower limb
* known severe psychiatric illness
* known malignancy, skin disease, infectious disease, severe cardiovascular disease, patients taking anti-coagulants
* enrolled in other studies
* refuse to temporarily discontinue concurrent treatment or intervention as pain management during the study period e.g. alternative medicine, physiotherapy, chiropractor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-06 (Actual); Primary Completion 2022-12-06 (Estimated); Study Completion 2023-09-06 (Estimated)

PRIMARY OUTCOMES:
Change of Pain Score | 3 different time points that include before the study (0 week), the mid term (12th week) and end of the study (24th weeks)
  The pain score in Numeric Rating Scale (0-10) for both groups of patients, which 0= no pain to 10=worst pain.

SECONDARY OUTCOMES:
Change of Endurance strength test of lower extremities | 3 different time points that include before the study (0 week), the mid term (12th week) and end of the study (24th weeks)
  For the test of lower extremities, study subjects will be asked to sit comfortably on a chair with the back straight. The arms are extended parallel to the trunk with the elbow and shoulder in 0° of flexion/extension, and each hand hold a dumbbell weighing 2.5kg. On receiving a signal from a metronome, subjects rise to a full standing position (body erect and straight), and at the next signal of the metronome, they return back to the initial seated position, maintaining arm extension. The pace of the metronome is 60 beats per minute and 90° of movement per second. The score is measured as the total number of stands executed correctly until the participant cannot keep up with the pace of the metronome.
Change of Endurance strength test of upper extremities | 3 different time points that include before the study (0 week), the mid term (12th week) and end of the study (24th weeks)
  For the test of upper extremities, you sit on the same chair, leaning back completely, extending the dominant arm parallel to the trunk with the elbow and shoulder in 0° of flexion/extension, and holding a dumbbell weighing 2.5kg. At the signal of the metronome, you bend the weight through a full range of elbow flexion. At the next signal of the metronome, you return to the initial position, keeping the back straight. The pace of the metronome is 60 beats per minute and 120° of movement per second. The score is measured as the total number of curls executed correctly until you cannot keep up with the pace of the metronome. This test is repeated on the other arm. The tests are approximately 5 to 10 minutes per patient.
Change of Brief pain inventory-Short Form (BPI) | 3 time points (0 week, 12th week and 24th week after obtaining consent)
  BPI measures clinical pain. It allows cases to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function. A scale of 0-10, 0=no interference and 10= completely interference.
Change of Hospital anxiety and depression scale (HADS) | 3 time points (0 week, 12th week and 24th week after obtaining consent)
  HADS determines the level of anxiety and depression that subjects are experiencing during the study period. It consists of 14 items scale of which 7 items relate to anxiety and 7 relate to depression. Each item is scored from 0-3 (0=normal; 3=worst) and a cut off point of 8/21 for either anxiety or depression.
Change of 36-item Short form Survey (SF-36) | 3 time points (0 week, 12th week and 24th week after obtaining consent)
  SF-36 measures health and mental status, which consists of 8 scaled scores. The 8 scaled scores are: vitality, physical functioning, bodily pain, general health perceptions, physical health functioning, emotional role functioning, social role functioning, & mental health. Each scale is directly transformed into a 0-100 scale [0=disability to 100=no disability].
Jenkins Sleep Evaluation Questionnaire (JSEQ) for sleep | 3 time points (0 week, 12th week and 24th week after obtaining consent)
  JSEQ evaluate the impact of therapies upon sleep problems. It is a 4 items questionnaire with a score of 0-5 for each item. A total score of 0= no sleep disturbance to 20 = highest sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Pik Yu Chen, RN, BSc, MSc, Principal Investigator — Pain Nurse (Registered Nurse)
Locations (1):
- Pain Management Centre (NTEC); PWH/ AHNH, Shatin, New Territories, Hong Kong